CLINICAL TRIAL: NCT02349659
Title: A Randomised Controlled Trial to Evaluate the Efficacy of the Spinal Modulation Axium® NeuroStimulator THerapy as a Treatment for Persistent INGuinal Pain Following Surgical Intervention: SMASHING
Brief Title: A Multi-Centre RCT of the Axium® Neurostimulator for the Treatment of Chronic Inguinal Pain Following Surgery
Acronym: SMASHING
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor withdrawn due to low inclusion rate
Sponsor: Maxima Medical Center (Other)
Responsible Party: Principal Investigator, Frederique Mol, drs., Maxima Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 24-SMI-2014
Record Dates: First submitted 2015-01-09; First posted 2015-01-29 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Chronic Inguinal Pain Refractory to Previous Surgical Intervention (Neurectomy)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conservative Medical Management (No Intervention): Continued medical management restricted to exclude interventional pain treatments
- Axium Group (Active Comparator): As the CMM group but also treated with Dorsal Root Ganglion stimulation using the Axium neurostimulator
  Interventions: Device: Implantation with the commercially available Axium neurostimulator

INTERVENTIONS:
Device: Implantation with the commercially available Axium neurostimulator
  Arms: Axium Group

SUMMARY:
24-SMI-2014 is a Randomised Controlled Trial with an optional one way cross-over comparing Conservative Medical Management (CMM) to treatment with the Axium neurostimulator + CMM. Subject population is chronic inguinal pain refractory to previous surgical intervention (neurectomy).

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 18 years old
2. Subject is able and willing to comply with the follow-up schedule and protocol
3. Chronic inguinal pain following Pfannenstiel Incision or Open Inguinal Hernia Repair for at least 6 months
4. Previously undergone neurectomy procedure as a treatment for chronic inguinal pain
5. Minimum daily average baseline pain rating of 5 out of 10 in the inguinal area on an 11-point NPRS
6. Subject is able to provide written informed consent
7. Meets of the inclusion criteria for the implantation of a neurostimulation system as set out by the Dutch Neuromodulation Society
8. Subject has been screened by a multi-disciplinary panel including the designated psychologist of the Máxima Medical Center and deemed suitable for implantation

Exclusion Criteria:

1. Female subject of childbearing potential is pregnant/nursing or plans to become pregnant during the course of the Trial
2. Escalating or changing pain condition within the past month as evidenced by investigator examination
3. Subject has had injection therapy or radiofrequency treatment of a target neural structure within the past 3 months
4. Subject currently has an active implantable device including implantable cardioverter defibrillator, pacemaker, spinal cord stimulator or intrathecal drug pump
5. Subject is unable to operate the device
6. Subjects currently has an active infection
7. Subject has participated in another clinical investigation within 30 days
8. Subject has a coagulation disorder or uses anticoagulants that, in the opinion of the investigator, precludes participation
9. Subject has a current or on going condition, which will probably require MRI investigation sometime in the following 2 years
10. Subject has had a spinal surgical procedure at or between vertebral levels T10-L2
11. Subject has been diagnosed with cancer in the past 2 years, except for skin malignancies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-12; Primary Completion 2017-07 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects experiencing ≥50% reduction in average daily pain intensity in the Axium Group as compared to the CMM only group using an eleven point (0-10) numerical pain rating scale (NPRS) | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Máxima Medisch Centrum, Eindhoven, Netherlands

REFERENCES:
- [Derived] Mol F, Scheltinga M, Roumen R, Wille F, Gultuna I, Kallewaard JW, Elzinga L, van de Minkelis J, Nijhuis H, Stronks DL, Huygen FJPM. Comparing the Efficacy of Dorsal Root Ganglion Stimulation With Conventional Medical Management in Patients With Chronic Postsurgical Inguinal Pain: Post Hoc Analyzed Results of the SMASHING Study. Neuromodulation. 2023 Dec;26(8):1788-1794. doi: 10.1016/j.neurom.2022.09.014. Epub 2022 Nov 29. PMID 36456417
- [Derived] Mol FMU, Roumen RM, Scheltinga MR. Comparing the efficacy of targeted spinal cord stimulation (SCS) of the dorsal root ganglion with conventional medical management (CMM) in patients with chronic post-surgical inguinal pain: the SMASHING trial. BMC Surg. 2018 Mar 27;18(1):18. doi: 10.1186/s12893-018-0349-8. PMID 29587729